CLINICAL TRIAL: NCT04584203
Title: Diastolic dYsfunctioN AssessMent in critICally Ill Patients: an Observational Prospective Multicentric Study.
Brief Title: Diastolic dYsfunctioN AssessMent in critICally Ill Patients
Acronym: DYNAMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: DYNAMIC
Record Dates: First submitted 2020-07-24; First posted 2020-10-12 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Critical Illness; Diastolic Dysfunction; Diastolic Heart Failure; Weaning Failure; Mechanical Ventilation Complication
MeSH Terms: conditions — Critical Illness; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bedside Echocardiography — All the intensivists performing the TTE in the involved centers fulfill the criteria of the American Society of Echocardiography and of the European Society of Intensive Care.
  Medicine to be considered as experts in critical care echocardiography. Each center performs the TTE evaluation by means of the ultrasound device available in the unit equipped with the tissue Doppler imaging program and a phased array transducer of 2.5 MHz and doppler signals is recorded along with the electrocardiogram.
  For the purpose of this study, the following TTE parameters are recorded from the apical 4-chamber view during each set of measurements:
Procedure: Spontaneuos breathing trial — The Spontaneous Breathing Trial will be performed accordingly to the clinical practice of the involved centers (a total support - including positive end-expiratory pressure plus pressure support equal or lower to 8 cmH20)
Diagnostic Test: Bedside Echocardiography_1 — Echocardiography performed within 24h from patient's admission - not optional
  Other Names: Baseline Echo_1
Diagnostic Test: Bedside Echocardiography_2 — Echocardiography performed within 12h from patient's spontaneous breathing trial - not optional
  Other Names: Echo_2
Diagnostic Test: Bedside Echocardiography_3 — Echocardiography performed at 60 +/- 12h from patient's admission - optional
  Other Names: Echo_3
Diagnostic Test: Bedside Echocardiography_4 — Echocardiography performed 24h after patient's estubation - optional
  Other Names: Echo_4

SUMMARY:
The role of the left ventricular diastolic function (LVDD) in the weaning failure from mechanical ventilation in unclear. Specifically, is unclear whether the outcome of the weaning process could be affected by a pre-existing LVDD (before ICU admission), or by the worsening of a chronic pattern, or by a de-novo LVDD presentation.

DETAILED DESCRIPTION:
Bedside echocardiography plays a critical diagnostic role in patients with heart failure, being other examinations (i.e., physical examination, electrocardiogram, and chest radiograph) unable to provide key information to discriminate between diastolic and systolic heart failure. Transthoracic echocardiography (TTE) can assess diastolic function by means of the doppler filling pattern, and can non-invasively measure intracardiac pressure at the bedside.

During sinus rhythm, diastolic flow shows the E and A waves, which reflects early diastolic filling and atrial contraction in the late diastole, respectively. Velocity of blood flow across the mitral valve depends on the trans-mitral pressure gradient; then, E-wave velocity is influenced both by the rate of early diastolic relaxation and by the left atrial pressure. Changes of the velocity pattern can suggest left ventricular diastolic function (LVDD) and prognosis, although mitral inflow patterns are highly susceptible to loading conditions (mainly left atrial pressure). LVDD is quite is a condition quite common in the population. A cross-sectional survey of over 2000 randomly selected Minnesota residents aged 45 years or older found an incidence of LVDD almost five times higher than LV systolic dysfunction (28% vs. 6%, respectively), which was a strong predictor of mortality (hazard ratio ranging from 8.3 for mild LVDD to 10.2 for at-least-moderate LVDD).

In a randomly recruited population sample (n = 539; 50.5% women; mean age, 52.5 years), the prevalence of the LVDD in those patients older than 50 y.o. was of about 50%5.

Doppler echocardiography could be a noninvasive tool for the detection of weaning-induced left ventricular filling pressure elevation. Transmitral flow can help measure peak Doppler velocities of E and A waves. E/A ratio has been proposed to estimate the left ventricular filling pressure. Tissue Doppler imaging can measure early diastolic mitral annular velocity (E'), which is a load-independent indicator of myocardial relaxation. The combination of tissue Doppler imaging and pulsed Doppler transmitral flow can allow the computation of the E/E' ratio, which is one of the best echocardiographic estimate of left ventricular filling pressure.

The role of LVDD in critically ill patients is probably greatly underestimated by intensivists, probably because in the past diastolic function was difficult to evaluate at the bedside6. The LVDD in intensive care unit (ICU) patients can affect the outcome of weaning from mechanical ventilation, especially in septic patients. In fact, cardiogenic pulmonary edema has been recognized as a highly incident cause of weaning failure. Unsuccessful weaning from mechanical ventilation occurs in approximately 20% of patients and is related to prolonged mechanical ventilation, length of stay in the intensive care unit, and increased morbidity and mortality. It has been proved that a spontaneous breathing trial (SBT) increases the left ventricular filling pressure, leading to cardiogenic pulmonary edema and impaired gas exchange.

However, studies focused on the impact of that medical condition on weaning showed conflicting results. Moreover, heterogeneous definitions and measurements of LVDD have been provided, associated to different form of SBTs. Furthermore, the majority carried out a cross-sectional assessment of the LVDD before and after the SBT, not including changes in the diastolic function during the ICU stay. All these variables limit the comparability and the clinical applications of these studies.

Moreover, LV diastolic function depends on myocardial relaxation, LV stiffness, and filling pressures, which are frequently impaired during the ICU stay (e.g., progression of the disease, volume resuscitation, positive end-expiratory pressure, administration of inotropes, vasopressors, etc). It is still uncertain whether the SBT failure could be affected by pre-existing conditions (i.e. a LVDD present at the ICU admission) or by a worsening of the cardiac function after the ICU admission.

As a matter of fact, the assessment of LVDD at the bedside is not routinely performed before the SBT and the role of the degree of the LVDD in still not defined. Moreover, it unclear whether the outcome of the weaning process could be affected by a pre-existing LVDD (before ICU admission), or by the worsening of a chronic pattern, or by a de-novo LVDD presentation.

ELIGIBILITY:
Inclusion criteria:

* Expected to be ventilated for >48 hours
* Age > 50

Exclusion criteria:

* Atrial fibrillation (at the admission or during ICU stay);
* Neuromuscular disorders

  •. Severe neurological events (traumatic or not) with GCS < 8 at admission
* Home ventilation prior to admission;
* Palliative intubation;
* Intubation for an indication to tracheostomy;
* Poor acoustic window (after the first assessment);
* Severe mitral and/or aortic valve stenosis or regurgitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to General ICU
Sampling Method: Non-Probability Sample
Enrollment: 297 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Spontaneous breathing trial failure | 6 hour after Spontaneous breathing trial end
  Patients admitted with LVDD
Spontaneous breathing trial failure | 6 hour after Spontaneous breathing trial end
  Patients worsening a pre-existing LVDD or developing a LVDD during the ICU stay.

SECONDARY OUTCOMES:
Prevalence of LVDD in critically ill patients | up to 3 weeks
  Echocardiography measurements
To assess the degree of the LVDD in critically ill patients | up to 3 weeks
  Echocardiography measurements
To correlate LVDD with clinical outcomes | up to 3 weeks
  Echocardiography measurements

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Messina, PhD, Principal Investigator — Humanitas Mirasole SpA
Locations (8):
- Italy (8):
  - Humanitas Research Hospital, Rozzano, Milano
  - Ospedale Ss. Trinità, Borgomanero, Novara
  - Careggi University Hospital, Florence, Tuscany
  - "Policlinico-San Marco", Catania
  - Azienda Ospedaliera di Perugia, Perugia
  - Grande Ospedale Metropolitano, Reggio Calabria
  - Policlinico Universitario A. Gemelli, Roma
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine

IPD SHARING:
Plan to Share IPD: Undecided
Raw data available from the PI, under reasonable reason

REFERENCES:
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Schmidt GA, Girard TD, Kress JP, Morris PE, Ouellette DR, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Truwit JD. Liberation From Mechanical Ventilation in Critically Ill Adults: Executive Summary of an Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline. Chest. 2017 Jan;151(1):160-165. doi: 10.1016/j.chest.2016.10.037. Epub 2016 Nov 3. PMID 27818329
- [Background] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740
- [Background] de Meirelles Almeida CA, Nedel WL, Morais VD, Boniatti MM, de Almeida-Filho OC. Diastolic dysfunction as a predictor of weaning failure: A systematic review and meta-analysis. J Crit Care. 2016 Aug;34:135-41. doi: 10.1016/j.jcrc.2016.03.007. Epub 2016 Mar 16. PMID 27067288
- [Background] Vignon P. Ventricular diastolic abnormalities in the critically ill. Curr Opin Crit Care. 2013 Jun;19(3):242-9. doi: 10.1097/MCC.0b013e32836091c3. PMID 23624639